CLINICAL TRIAL: NCT03616314
Title: Effects of Early Stepping Verticalization With or Without FES Compared to Conventional Physiotherapy on the Occurrence of Critical Illness Polyneuropathy in Patients Affected by Acquired Brain Injury: a Retrospective Study
Brief Title: Effects of Early Stepping Verticalization + FES on CIP
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: Erigo/FES critical illness
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Critical Illness Polyneuropathy; Acquired Brain Injury
MeSH Terms: conditions — Polyneuropathies; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- stepping verticalization: in ICU they received conventional physiotherapy + stepping verticalization sessions with Erigo
  Interventions: Device: stepping verticalization
- stepping verticalization + FES: in ICU they received conventional physiotherapy + stepping verticalization sessions with FES using ErigoPro
  Interventions: Device: stepping verticalization plus functional electrical stimulation
- conventional physiotherapy: in ICU they received only conventional physiotherapy
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Device: stepping verticalization plus functional electrical stimulation — patients hospitalized in ICU are rehabilitated using 30 minutes/day of conventional physiotherapy + 30 minutes/day of verticalization using a tilt table with an integrated robotic stepping device synchronized with an electrical stimulation of the lower limbs muscles
  Groups: stepping verticalization + FES
Device: stepping verticalization — patients receive 30 minutes/day of conventional physiotherapy + 30 minutes7day of verticalization using a tilt table with a robotic stepping device
  Groups: stepping verticalization
Other: conventional physiotherapy — patients are treated only with 60 minutes/day of conventional physiotherapy
  Groups: conventional physiotherapy

SUMMARY:
Background: Intensive Care Unit (ICU) survivors often develop an acquired weakness due to a Critical Illness Polyneuropathy (CIP). Early mobilization in ICU, by reducing the bed rest and decreasing the oxidative stress, was shown to represent a valid preventive option.

Purpose: To evaluate whether ICU sessions of stepping verticalization associated with Functional Electrical Stimulation (FES) of the lower limbs are able to reduce the occurrence of CIP in Acquired Brain Injured (ABI) patients.

Methods: all the ABI patients admitted in our Neurorehabilitation Unit from our ICU were retrospectively evaluated. Patients affected by previous peripheral neuropathy, diabetes, cancer, alcoholism, viral hepatitis, AIDS and autoimmune diseases were excluded. They were divided into 3 groups according to the rehabilitation strategy received in ICU: group 1 received conventional physiotherapy + stepping verticalization sessions with Erigo® (Hocoma, Switzerland); group 2 received conventional physiotherapy + stepping verticalization sessions with FES using ErigoPro®; group 3 received only conventional physiotherapy. As for internal protocol, all patients started rehabilitation in the first week from the ABI and performed 60 minutes/day of rehabilitation, 5 days/week. Primary outcome was the evidence of CIP at Neurorehabilitation admission (=ICU discharge), according to neurophysiological criteria. Secondary outcomes were the strength impairment at Neurorehabilitation discharge, measured by the total Motricity Index score and the Functional Ambulation Classification (FAC) score, assessing quality of gait.

ELIGIBILITY:
Inclusion Criteria:

* arriving directly from our acute care facility
* hospitalized in ICU due to an acute brain injury

Exclusion Criteria:

* previous peripheral neuropathies
* diabetes
* cancer
* alcoholism
* viral hepatitis
* AIDS
* autoimmune diseases
* absence of clinical or neurophysiological informations at data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in ICU and transferred in Neurorehab after an acute brain injury
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
CIP occurrence | at enrollment
  Presence of critical illness polyneuropathy at the end of ICU stay

SECONDARY OUTCOMES:
motricity index | at enrollment
  total motricity index score (4 limbs) at neurorehabilitation discharge. Score goes from 0 (no movement in any limb) to 400 (full strength in alla limbs)
Functional Ambulation Classification (FAC) | at enrollment
  Functional Ambulation Classification score at neurorehabilitation discharge. Scale goes from 0 (no ambulation) to 5 (independent ambulation)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona Moriggia Pelascini, Gravedona, CO, Italy